CLINICAL TRIAL: NCT05342649
Title: "Effect of Two Methods of Soft Tissue Augmentation for Socket Closure on Soft Tissue Landmarks and Ridge Dimensions- Results From Software-based Analysis of Clinical Data"
Brief Title: Effect of Two Methods of Soft Tissue Augmentation for Socket Closure on Soft Tissue Landmarks and Ridge Dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/1/2017
Record Dates: First submitted 2022-04-08; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main treatment group (Experimental): soft tissue closure of extraction sockets was done by pediculated connective tissue grafts (P-CTG)
  Interventions: Procedure: P-CTG
- Control group (Active Comparator): soft tissue closure of extraction sockets was done by connective tissue grafts (CTG)
  Interventions: Procedure: CTG

INTERVENTIONS:
Procedure: P-CTG — soft tissue closure of extraction sockets was done by pediculated connective tissue grafts (P-CTG)
  Other Names: Experimental group
  Arms: Main treatment group
Procedure: CTG — soft tissue closure of extraction sockets was done by connective tissue grafts (CTG)
  Other Names: Control group
  Arms: Control group

SUMMARY:
To evaluate the effect of Connective Tissue Graft and Pediculated-Connective Tissue Graft for extraction socket closure on soft tissue landmarks and ridge dimensions.

DETAILED DESCRIPTION:
45 subjects were randomized into two groups Experimental: Main treatment group P-CTG group Active Comparator: Control group CTG group.

ELIGIBILITY:
Inclusion Criteria:

* Based on the Extraction Defect Sounding(EDS) Classification given by Caplanis et al,

  1. Systemically healthy subjects within the age group of 20-50years
  2. with extraction defect type 2 and type 3 were included in this study

Exclusion Criteria:

1. Medically compromised patients
2. Subjects who underwent radiotherapy or chemotherapy and
3. Smokers

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
BL Gain | Baseline to 6 months
  The displacement from the baseline to 6-months in BL dimensions was calculated and was described as BL gain.
Total displacement (TD) | Baseline to 6 months
  The total displacement (TD) from the baseline to 6-months in MD dimensions was calculated and was described as TD gain.
Angle of Displacement (AOD) | Baseline to 6 months
  The Angle of Displacement (AOD)) from the baseline to 6-months in MD dimensions was calculated and was described as AOD Change.

CONTACTS AND LOCATIONS:
Overall Officials: Bhagyasree Medisetty, MDS, Principal Investigator — SVS Institute of Dental Sciences
Locations (1):
- SVS Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No